CLINICAL TRIAL: NCT05458102
Title: A Phase 1, Open-label, Multicohort Study to Evaluate the Impact of Inhibitors and Inducers of Cytochrome P450 Enzyme (CYP)3A and/or P-glycoprotein (P-gp) on the Pharmacokinetics (PK) of Vesatolimod (VES) in Virologically Suppressed Adults With HIV-1 on Antiretroviral Therapy (ART)
Brief Title: Drug-Drug Interaction Study of Vesatolimod in Adults With HIV-1 Who Have Very Low or Undetectable Virus Levels
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision to change the clinical development plan of this molecule. This decision is not based on efficacy or safety concerns.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-382-1587
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Human Immunodeficiency Virus Type 1 (HIV-1) Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — vesatolimod; Cobicistat; Voriconazole; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Vesatolimod + Cobicistat + Voriconazole (Experimental): Participants will receive a single dose of vesatolimod (VES) 2 mg on Day 1 of Period 1. In Period 2, participants will receive cobicistat (COBI) 150 mg once daily on Days 1 to 5 along with a single dose of VES 2 mg on Day 2. In Period 3, participants will receive a loading dose of voriconazole (VOR) 400 mg twice daily on Day 1, then VOR 200 mg twice daily on Days 2 to 6, and a single dose of VES 2 mg in the morning on Day 3. There will be a washout period of 7 to 14 days between treatments in Period 1 Day 1 and Period 2 Day 1 and a washout period of 14 to 21 days between treatments in Period 2 Day 5 and Period 3 Day 1.
  Interventions: Drug: Vesatolimod; Drug: Cobicistat; Drug: Voriconazole
- Cohort 2: Vesatolimod + Rifabutin (Experimental): Participants will receive a single dose of VES 6 mg on Day 1. In Period 2, participants will receive Rifabutin (RFB) 300 mg once daily on Days 1 to 9 along with a single dose of VES 6 mg on Day 6. There will be a washout period of 7 to 14 days between treatments in Period 1 Day 1 and Period 2 Day 1.
  Interventions: Drug: Vesatolimod; Drug: Rifabutin

INTERVENTIONS:
Drug: Vesatolimod — Administered orally
  Other Names: GS-9620
Drug: Cobicistat — Administered orally
  Other Names: Tybost®
  Arms: Cohort 1: Vesatolimod + Cobicistat + Voriconazole
Drug: Voriconazole — Administered orally
  Other Names: Vfend®
  Arms: Cohort 1: Vesatolimod + Cobicistat + Voriconazole
Drug: Rifabutin — Administered orally
  Other Names: Mycobutin®
  Arms: Cohort 2: Vesatolimod + Rifabutin

SUMMARY:
The goal of this clinical study is to learn more about the impact of cobicistat (COBI) (P-glycoprotein (P-gp), breast cancer resistance protein (BCRP), and strong cytochrome P450 enzyme [CYP]3A inhibitor), voriconazole (VOR) (strong CYP3A inhibitor), and rifabutin (RFB) (moderate CYP3A inducer) on the study drug, vesatolimod (VES), in people with HIV-1 on antiretroviral therapy (ART).

ELIGIBILITY:
Key Inclusion Criteria:

* On an antiretroviral therapy (ART) regimen for at least 6 consecutive months, with no change in the ART regimen within 2 months prior to screening. Permitted ARTs are as follows:

  * Cohort 1: A regimen of (bictegravir [BIC], dolutegravir [DTG], raltegravir [RAL], or doravirine [DOR]) plus Nucleoside Reverse Transcriptase Inhibitors (NRTIs). Examples of acceptable regimens include BIC/emtricitabine/tenofovir, DTG/ abacavir (ABC)/3TC, DTG/3TC, DTG + emtricitabine/tenofovir, or DOR/3TC/tenofovir
  * Cohort 2: A DTG-based regimen is required (DTG/ABC/3TC), (DTG/3TC), or (DTG + NRTIs)
* Plasma HIV-1 RNA levels less than 50 copies/mL at screening
* Have normal hematologic function with an absolute neutrophil count greater than or equal to 1.5 × 10^9/L, platelets greater than or equal to 150 × 10^9/L; hemoglobin greater than or equal to 10.5 g/dL for females and greater than or equal to 11.5 g/dL for males
* Clusters of differentiation (CD) 4 T cell count greater than or equal to 350 cells/μL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x upper limit of normal (ULN) and total bilirubin less than or equal to 1.5 mg/dL, or normal direct bilirubin and creatinine less than or equal to 1.25 x ULN
* Have a calculated creatinine clearance (CLcr) of at least 60 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at screening and upon admission
* Individuals assigned female at birth and of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception
* Must be willing and able to comply with all study requirements and available to complete the study schedule of assessments
* In the judgment of the investigator, be in good general health, based on review of the results from a screening visit

Key Exclusion Criteria:

* Have received any study drug within 30 days prior to study dosing
* Participation in any other clinical study (including observation studies) without prior approval from the sponsor is prohibited while participating in this study
* Have current alcohol or substance abuse judged by the investigator to potentially interfere with individual compliance or individual safety, or a positive drug or alcohol test at screening or baseline
* No Evidence of chronic hepatitis B virus (HBV) infection (defined as positive hepatitis B surface antigen [HBsAg] and/or positive HBV core antibody with positive reflex HBV DNA polymerase chain reaction (PCR)). Note: positive HBV core antibody with negative reflex HBV DNA PCR results are acceptable
* No Evidence of active hepatitis C virus (HCV) infection (defined as positive hepatitis C antibody and HCV RNA above lower limit of quantitation). Note: positive anti-HCV antibody and negative HCV PCR results are acceptable
* Acute febrile illness within 35 days prior to Day 1
* Have been treated with systemic steroids, immunosuppressant therapies, or chemotherapeutic agents within 3 months prior to screening or is expected to receive these agents during the study
* Received any vaccine or immunomodulatory medication within 4 weeks prior to screening. Elective vaccination (eg, flu shot, hepatitis A or B vaccine) during the course of the study will require prior approval from the sponsor

  * Coronavirus disease of 2019 (COVID-19) vaccinations are allowed, with the requirement that they should not be administered within 7 ± 2 days of receiving VES
* Have a history of any of the following:

  * Significant serious skin disease, such as but not limited to rash, food allergy, eczema, psoriasis, or urticaria
  * Significant drug sensitivity or drug allergy (such as anaphylaxis or hepatoxicity)
  * Known hypersensitivity to the study drugs, their metabolites, or to formulation excipients
  * Autoimmune disease
  * Significant cardiac disease or a family history of long QT syndrome, or unexplained death in an otherwise healthy individual between the ages of 1 and 30 years
  * Syncope, palpitations, or unexplained dizziness
  * Implanted defibrillator or pacemaker
  * Liver disease, including Gilbert syndrome
  * Severe peptic ulcer disease requiring prolonged (≥ 6 months) medical treatment
  * Medical or surgical treatment that permanently altered gastric absorption (eg, gastric or intestinal surgery). A history of cholecystectomy is not exclusionary
* Have any serious or active medical or psychiatric illness (including depression) that, in the opinion of the investigator, would interfere with individual treatment, assessment, or compliance with the protocol
* For Cohort 1, individuals with CYP2C19 genotype of CYP2C19*2/*2, CYP2C19*2/*3, or CYP2C19*3/*3

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - Collaborative Neuroscience Research, LLC., Long Beach, California
  - Clinical Pharmacology of Miami, LLC., Miami, Florida
  - Advanced Pharma, CR, LLC., Miami, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Hassman Research Institute, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng Y, Wire M, Omange RW, deVries CR, Zhang L, Chen B, Huang SSY, Cruz K, Hassman H, Osiyemi O, Rondon JC, Lim D, West S, Wen A, Wallin JJ, SenGupta D, Cai Y. The Effects of Cobicistat and Voriconazole on the Safety, Pharmacokinetics, and Pharmacodynamics of the TLR7 Agonist Vesatolimod in People with HIV. Infect Dis Ther. 2025 Nov;14(11):2535-2549. doi: 10.1007/s40121-025-01227-x. Epub 2025 Sep 15. PMID 40952649
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-382-1587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 59 participants were screened.
Groups:
- Cohort 1: Vesatolimod + Cobicistat + Voriconazole: Participants received a single dose of vesatolimod (VES) 2 mg on Day 1 of Period 1. In Period 2, participants received cobicistat (COBI) 150 mg once daily on Days 1 to 5 along with a single dose of VES 2 mg on Day 2. In Period 3, participants received a loading dose of voriconazole (VOR) 400 mg twice daily on Day 1, then VOR 200 mg twice daily on Days 2 to 6, and a single dose of VES 2 mg in the morning on Day 3. There was a washout period of 7 to 14 days between treatments in Period 1 Day 1 and Period 2 Day 1 and a washout period of 14 to 21 days between treatments in Period 2 Day 5 and Period 3 Day 1.
- Cohort 2: Vesatolimod + Rifabutin: Participants received a single dose of VES 6 mg on Day 1. In Period 2, participants received Rifabutin (RFB) 300 mg once daily on Days 1 to 9 along with a single dose of VES 6 mg on Day 6. There was a washout period of 7 to 14 days between treatments in Period 1 Day 1 and Period 2 Day 1.
Period: Overall Study
Arm/Group | Cohort 1: Vesatolimod + Cobicistat + Voriconazole | Cohort 2: Vesatolimod + Rifabutin
Started | 16 | 2
Completed | 11 | 2
Not Completed | 5 | 0
Not completed — Withdrew consent | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Enrolled but never treated | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Vesatolimod + Cobicistat + Voriconazole | Cohort 2: Vesatolimod + Rifabutin | Total
Number analyzed (Participants) | 15 | 2 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 2 | 16
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14.5) | 45 (14.8) | 47 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data for Cohort 2 are not reported due to participants' confidentiality reasons as there were only 2 participants in this cohort.
  Participants
    number analyzed (Participants) | 15 | 0 | 15
    Female | 2 | 0 | 2
    Male | 13 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data for Cohort 2 are not reported due to participants' confidentiality reasons as there were only 2 participants in this cohort.
  Participants
    number analyzed (Participants) | 15 | 0 | 15
    Hispanic or Latino | 3 | 0 | 3
    Not Hispanic or Latino | 12 | 0 | 12
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data for Cohort 2 are not reported due to participants' confidentiality reasons as there were only 2 participants in this cohort.
  Participants
    number analyzed (Participants) | 15 | 0 | 15
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 10 | 0 | 10
    White | 2 | 0 | 2
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter : AUClast of Vesatolimod (VES)
Description: AUClast is defined as an area under the concentration versus time curve from time zero to the last quantifiable concentration.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose for Cohort 1 on Period 1 Day 1, Period 2 Day 2, and Period 3 Day 3; and for Cohort 2 on Period 1 Day 1 and Period 2 Day 6
Population: The VES PK Analysis Set included participants who received at least 1 dose of VES and had at least 1 nonmissing PK concentration value.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Groups:
- Cohort 1: Vesatolimod 2 mg: Participants received a single dose of VES 2 mg on Day 1 of Period 1.
- Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg: Participants received COBI 150 mg once daily on Days 1 to 5 along with a single dose of VES 2 mg on Day 2 in Period 2.
- Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg: Participants received VOR 200 mg twice daily on Days 2 to 6, and a single dose of VES 2 mg in the morning on Day 3 in Period 3.
- Cohort 2: Vesatolimod 6 mg: Participants received a single dose of VES 6 mg on Day 1 in Period 1.
- Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg: Participants received RFB 300 mg once daily on Days 1 to 9 along with a single dose of VES 6 mg on Day 6 in Period 2.
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 15 | 13 | 11 | 2 | 2
h*pg/mL | 13500 (9500) | 61900 (35400) | 14600 (11000) | 16400 (17900) | 86300 (16000)
Statistical Analysis 1: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg; Test type: Other; Geometric Least-squares Mean Ratio = 560, 90% CI 2-sided [414 to 757] — Parametric (normal theory) mixed-effects ANOVA model was fitted to the natural log-transformed values of the PK parameter under evaluation
Statistical Analysis 2: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg; Test type: Other; Geometric Least-squares Mean Ratio = 137, 90% CI 2-sided [99.5 to 189] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: PK Parameter : AUCinf of VES
Description: AUCinf is defined as an area under the concentration versus time curve extrapolated to infinite time, calculated as AUClast + (Clast/Lambda z).
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: Participants in the VES PK Analysis Set with available data were analyzed. Data for Cohort 2 Vesatolimod 6mg are not reported due to participant's confidentiality reasons as there was only 1 participant in this cohort.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 13 | 12 | 10 | 0 | 2
h*pg/mL | 17600 (9220) | 68000 (36600) | 17800 (11600) |  | 88000 (16800)
Statistical Analysis 1: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg; Test type: Other; Geometric Least-squares Mean Ratio = 433, 90% CI 2-sided [347 to 540] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg; Test type: Other; Geometric Least-squares Mean Ratio = 118, 90% CI 2-sided [93.5 to 150] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: PK Parameter : Cmax of VES
Description: Cmax is defined as the maximum observed concentration of drug.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: Participants in the VES PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 15 | 13 | 11 | 2 | 2
pg/mL | 1130 (1020) | 6930 (4650) | 1020 (895) | 944 (928) | 22200 (7780)
Statistical Analysis 1: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg; Test type: Other; Geometric Least-squares Mean Ratio = 752, 90% CI 2-sided [525 to 1080] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg; Test type: Other; Geometric Least-squares Mean Ratio = 118, 90% CI 2-sided [80.3 to 172] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: PK Parameter : %AUCexp of VES
Description: %AUCexp is defined as the percentage of AUC extrapolated between AUClast and AUCinf, calculated as ([AUCinf-AUClast]/AUCinf)*100.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of AUCexp
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 13 | 12 | 10 | 0 | 2
percentage of AUCexp | 14.6 (6.97) | 6.16 (3.91) | 14.7 (6.75) |  | 1.92 (0.602)

5. Primary Outcome: PK Parameter : Tmax of VES
Description: Tmax is defined as the time (observed time point) of Cmax.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: Participants in the VES PK Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 15 | 13 | 11 | 2 | 2
hours | 3.03 [1.50 to 6.00] | 1.52 [1.50 to 2.48] | 2.50 [1.00 to 3.10] | 5.13 [4.18 to 6.07] | 1.28 [1.05 to 1.50]
Statistical Analysis 1: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg; Test type: Other; Geometric Least-squares Mean Ratio = 68.5, 90% CI 2-sided [45.5 to 103] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg; Test type: Other; Geometric Least-squares Mean Ratio = 65.4, 90% CI 2-sided [42.5 to 101] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: PK Parameter : Clast of VES
Description: Clast is defined as the last observed quantifiable concentration of the drug.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: Participants in the VES PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 15 | 13 | 11 | 2 | 2
pg/mL | 84.2 (19.4) | 103 (42.2) | 74.2 (17.4) | 75.9 (30.5) | 74.3 (27.2)

7. Primary Outcome: PK Parameter : Tlast of VES
Description: Tlast is defined as the time (observed time point) of Clast.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: Participants in the VES PK Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 15 | 13 | 11 | 2 | 2
hours | 48.0 [24.1 to 72.0] | 72.0 [71.7 to 96.0] | 48.0 [24.3 to 96.0] | 59.8 [24.0 to 95.5] | 72.0 [72.0 to 72.0]

8. Primary Outcome: PK Parameter : Lambda z of VES
Description: Lambda z is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log concentration of drug versus time curve of the drug.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: per hour
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 14 | 12 | 11 | 0 | 2
per hour | 0.0381 [0.0310 to 0.0528] | 0.0310 [0.0252 to 0.0425] | 0.0321 [0.0241 to 0.0561] |  | 0.0442 [0.0400 to 0.0485]

9. Primary Outcome: PK Parameter : t1/2 of VES
Description: t1/2 is defined as the terminal elimination half-life.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 14 | 12 | 11 | 0 | 2
hours | 18.4 [13.1 to 22.3] | 22.4 [16.7 to 27.6] | 21.6 [12.4 to 28.7] |  | 15.8 [14.3 to 17.4]
Statistical Analysis 1: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg; Test type: Other; Geometric Least-squares Mean Ratio = 120, 90% CI 2-sided [104 to 138] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1: Vesatolimod 2 mg vs Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg; Test type: Other; Geometric Least-squares Mean Ratio = 111, 90% CI 2-sided [95.4 to 128] — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: PK Parameter : CL/F of VES
Description: CL/F is defined as an apparent oral clearance.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 13 | 12 | 10 | 0 | 2
L/h | 156 (92.9) | 42.4 (28.5) | 176 (137) |  | 69.4 (13.3)

11. Primary Outcome: PK Parameter : Vz/F of VES
Description: Vz/F is defined as an apparent volume of distribution of the drug.
  Cohort 1 Period 1 Day 1: Day 1 from Baseline; Cohort 1 Period 2 Day 2: Up to Day 17 from Baseline; Cohort 1 Period 3 Day 3: Up to Day 44 from Baseline; Cohort 2 Period 1 Day 1: Day 1 from Baseline; Cohort 2 Period 2 Day 6: Up to Day 21 from Baseline.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 13 | 12 | 10 | 0 | 2
L | 3480 (1530) | 1320 (1100) | 4330 (2220) |  | 1560 (86.7)

12. Primary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a study drug that does not necessarily have a causal relationship with the treatment. An AE can, therefore, be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug. Adverse events may also include pretreatment or posttreatment complications that occur as a result of protocol-specified procedures, or special situations. TEAES included all AEs began on or after the study drug start date.
Time Frame: First dose date up to last dose date plus 30 days (up to 77 days for Cohort 1, and up to 54 days for Cohort 2)
Population: Participants in Safety Analysis Set were analyzed. Per planned analysis, the data for adverse events were summarized by study treatments administered in Cohorts 1 and 2 per period.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1: Cobicistat 150 mg: Participants received COBI 150 mg once daily on Days 1 to 5 in Period 2.
- Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg: Participants received COBI 150 mg once along with a single dose of VES 2 mg on Day 2 in Period 2.
- Cohort 1: Voriconazole 400 mg: Participants received a loading dose of VOR 400 mg twice daily on Day 1 in Period 3.
- Cohort 1: Voriconazole 200 mg: Participants received VOR 200 mg twice daily on Days 2 to 6 in Period 3.
- Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg: Participants received VOR 200 mg twice along with a single dose of VES 2 mg on Day 3 in Period 3.
- Cohort 2: Rifabutin 300 mg: Participants received RFB 300 mg once daily on Days 1 to 9 in Period 2.
- Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg: Participants received RFB 300 mg once along with a single dose of VES 6 mg on Day 6 in Period 2.
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Voriconazole 400 mg | Cohort 1: Voriconazole 200 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Rifabutin 300 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 15 | 13 | 13 | 11 | 11 | 11 | 2 | 2 | 2
percentage of participants | 13.3 | 38.5 | 0 | 36.4 | 9.1 | 9.1 | 0 | 50.0 | 50.0

13. Primary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 toxicity grade from predose at any time postdose. Data for participants with post baseline toxicity grade 1 or higher is reported.
Time Frame: First dose date up to last dose date plus 30 days (up to 77 days for Cohort 1, and up to 54 days for Cohort 2)
Population: Participants in Safety Analysis Set with available data were analyzed. Per planned analysis, the data for adverse events were summarized by study treatments administered in Cohorts 1 and 2 per period.
Measure: Number; unit: percentage of participants
Groups:
- Vesatolimod 2 mg + Cobicistat 150 mg: Participants received COBI 150 mg once along with a single dose of VES 2 mg on Day 2 in Period 2.
- Vesatolimod 2 mg + Voriconazole 200 mg: Participants received VOR 200 mg twice along with a single dose of VES 2 mg on Day 3 in Period 3.
- Vesatolimod 6 mg + Rifabutin 300 mg: Participants received RFB 300 mg once along with a single dose of VES 6 mg on Day 6 in Period 2.
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Cobicistat 150 mg | Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Voriconazole 400 mg | Cohort 1: Voriconazole 200 mg | Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 2: Vesatolimod 6 mg | Cohort 2: Rifabutin 300 mg | Vesatolimod 6 mg + Rifabutin 300 mg
Number analyzed (Participants) | 14 | 13 | 0 | 0 | 11 | 0 | 2 | 2 | 0
percentage of participants | 35.7 | 53.8 |  |  | 63.6 |  | 50.0 | 100.0 |

ADVERSE EVENTS:
Time Frame: Adverse Events and All-cause mortality: Up to 77 days for Cohort 1 and up to 54 days for Cohort 2
Description: All-cause mortality: All Enrolled Analysis Set included all participants who received study participant identification number in study after screening. Cohort 1: No treatment group is reported for 1 participant who was enrolled but never treated.
  Adverse Events: Safety Analysis Set included all participants who took at least 1 dose of study drug. Per planned analysis, Adverse Events/All-cause mortality were summarized by study treatments administered in Cohort 1 and Cohort 2 per period.
Groups:
- Cohort 1: No Treatment: Participant was enrolled but was not dosed.
Arm/Group | Cohort 1: Vesatolimod 2 mg | Cohort 1: Cobicistat 150 mg | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg | Cohort 1: Voriconazole 400 mg | Cohort 1: Voriconazole 200 mg | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg | Cohort 1: No Treatment | Cohort 2: Vesatolimod 6 mg | Cohort 2: Rifabutin 300 mg | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/13 | 0/11 | 0/11 | 0/11 | 0/1 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/13 | 0/11 | 0/11 | 0/11 | 0/0 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/15 | 5/13 | 0/13 | 4/11 | 1/11 | 1/11 | 0/0 | 0/2 | 1/2 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Vesatolimod 2 mg (N=15) | Cohort 1: Cobicistat 150 mg (N=13) | Cohort 1: Vesatolimod 2 mg + Cobicistat 150 mg (N=13) | Cohort 1: Voriconazole 400 mg (N=11) | Cohort 1: Voriconazole 200 mg (N=11) | Cohort 1: Vesatolimod 2 mg + Voriconazole 200 mg (N=11) | Cohort 1: No Treatment (N=0) | Cohort 2: Vesatolimod 6 mg (N=2) | Cohort 2: Rifabutin 300 mg (N=2) | Cohort 2: Vesatolimod 6 mg + Rifabutin 300 mg (N=2)
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT05458102/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT05458102/SAP_001.pdf